CLINICAL TRIAL: NCT03163823
Title: A Randomized Controlled Trial of an iPad for Patient Communication During Mechanical Ventilation
Brief Title: CTSI-iPad for Vented Patient Communication
Acronym: iPad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Marquette University (Other)
Responsible Party: Principal Investigator, Rahul Nanchal, Associate Professor of Medicine and Director of the Medical Intensive Care Unit, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 27533; 9665310 (Other Grant/Funding Number: CTSI of Southeast Wisconsin)
Record Dates: First submitted 2017-03-09; First posted 2017-05-23 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Communication (Placebo Comparator): Standard of Care communication styles will be used. Patients will receive the standard communication protocol identified by the hospital.
  Interventions: Other: Standard of Care
- iPad with Speech App (Experimental): Use of application Proloquo2Go on iPad device. The application being used is called Proloquo2Go which is the intervention portion. The iPad is the device used to access the application.
  Interventions: Other: Proloquo2Go

INTERVENTIONS:
Other: Proloquo2Go — Use of communication application Proloquo2Go modified for the ICU setting on an iPad device
  Arms: iPad with Speech App
Other: Standard of Care — Standard of Care communication methods
  Arms: Standard Communication

SUMMARY:
This study will enroll 75 mechanically vented adults in the ICU to compare self-reported ease of communication, patient satisfaction, and patient anxiety and frustration levels between a group using a communication application on an iPad and a group using standard methods of communication while mechanically vented.

DETAILED DESCRIPTION:
The Investigators will randomize patients to either an iPad application available for communication or usual care. An existing iPad communication application (Proloquo2Go) that allows picture or text to voice communication was tailored to needs of adult mechanically ventilated (MV) patient. In the tailored application, common messages for an adult MV population are depicted on picture tiles organized into folders. When patients touch a picture tile either additional message options appear or a phrase or word is spoken by the device. Access to a pop-up keyboard on each screen allows patients to easily type unique text to voice messages.

Intervention: Patients will be randomized to either an iPad with the tailored communication application or usual care. Patients randomized to the iPad group will be given a brief introduction to the communication application and then will be asked to communicate four messages to verify understanding. Patients who are unable to successfully use the iPad with the initial introduction will remain in the study. Research staff will continue to assist the patient daily and a speech language pathologist will be consulted to facilitate the patients ability to use the device. The iPad will remain at the bedside to be used for communication as desired for the remainder of the time the patient is on the ventilator. A manual providing instruction for the iPad and application operation will be at the bedside of all patients randomized to the intervention group. Research staff will visit patients daily to assist with any problems encountered and will also be available by phone to assist as needed. Although patients will be encouraged to use the iPad for communication, use of other strategies or tools will not be restricted.

ELIGIBILITY:
Inclusion Criteria:

1. Sufficient motor and visual function to allow use of touch screen
2. Mechanically ventilated
3. Awake and able to participate in informed consent discussion

Exclusion Criteria:

1. Non-English Speaking
2. Receiving ventilator support prior to admission.
3. Delirium present in the last 24 hours
4. Tracheostomy
5. Structural Neurological Injury (such as stroke or traumatic brain injury)
6. Coma
7. Deep Sedation (Richmond Agitation Scale > -2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Ease of Communication | 30 Days
  Patient self-reported ease of communication during mechanical ventilation measured using a Likert scale

SECONDARY OUTCOMES:
Patient Anxiety | 30 Days
  Patient Anxiety while Mechanically Ventilated in an ICU measured by VAS anxiety
Patient Satisfaction | 30 Days
  Mechanically ventilated ICU patient satisfaction with device measured using a Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Nanchal, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share.